CLINICAL TRIAL: NCT04576234
Title: Comparative Study Between the Effect of Intermittent Enteral Feeding by Syringe Pump and Hospital Blended Enteral Feeding by Feeding Bag on Complications and Nutritional Status Among ICU Patients.
Brief Title: Comparative Study Between Two Routes of Enteral Feeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarah Asmaa (Other)
Responsible Party: Sponsor-Investigator, Sarah Asmaa, clinical professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: enteral feeding; sasmaa (Registry Identifier: assiut university); Mostafa Samy (Registry Identifier: assiut university)
Record Dates: First submitted 2020-08-29; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Complication
Keywords: intermittent enteral feeding; hospital blended feeding; complications; nutritional status

STUDY DESIGN:
Intervention Model Description: After getting ethical clearance; patients were enrolled in the study, patients were selected based on the inclusion and exclusion criteria. Following an initial assessment, the patients were assigned to one of the two groups by block randomization.
  Both groups received 3000 ml of feed per day and the same formula per day which was 30-35ml/kg of water, 0.8 g/kg of protein and 2000 kcal of calories for females and 2500 Kcal for males. The only manipulation was in the flow rate and the device which the feed was administred.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intermittent entral feeding group (Experimental): Intermittent enteral feeding group recieved intermittent feeding as the feed was given over a 24 hour period with intervals of rest (e.g. three hours feeding two hours rest) by using syringe pump and Feeds were administered according to guidelines as the head of the patient's bed was elevated at least 30 degrees from the horizontal before initiating feeding, the feeding schedule was started at a rate of 50 ml/hr in adults to promote tolerance,the administration rate of isotonic formulas increased in 20-25 ml/hr increments every eight hours until the desired rate was achieved, the tube was flushed regularly with 20 to 30 ml of warm water every four hours during continuous feeding and before and after intermittent feeding and medication administration, the gastric residual volume was checked every 4-6 hr routinely
  Interventions: Dietary Supplement: entral feeding
- , feeding bag group (Experimental): Feeding bag group received hospital blended formual which was 300 ml of feeds every 2hrs with 4hrs rest at night and given in 10 minutes with following the same guidelines in the intermittent enteral feeding group
  Interventions: Dietary Supplement: entral feeding

INTERVENTIONS:
Dietary Supplement: entral feeding — Intermittent enteral feeding group recieved intermittent feeding as the feed was given over a 24 hour period with intervals of rest (e.g. three hours feeding two hours rest)

SUMMARY:
The study assess, evaluate and compare the efficacy of two methods of enteral feeding on complications and nutritional status among ICU patients.

The study had utilized two methods of enteral feeding consisted of intermittent enteral feeding by syringe pump and hospital blended enteral feeding by feeding bag and assess the patient before and after feeding for 10 days by using three tools help to monitor hemodynamic parameters, GIT system assessment and laboratory findings assessment which help to evaluate nutritional status and complications. The results showed that the complications in the intermittent enteral feeding group were lower than those in feeding bag group.

DETAILED DESCRIPTION:
Introduction Enteral nutritional support refers to the provision of calories, protein, electrolytes, vitamins, minerals, trace elements, and fluids via the gastrointestinal route. Enteral feeding is indicated for patients with a functional gastrointestinal tract whose oral nutritional intake is insufficient to meet estimated needs .

Enteral nutrition therapy has a number of advantages over par-enteral nutrition in the management of patients requiring nutritional support. Enteral nutrition aids in the preservation of gastrointestinal function by the provision of enteral nutrients and is easier, safer and less costly to administer .

However, despite these relative advantages, the delivery of safe and effective enteral nutrition therapy may still present challenges for families and caregivers in terms of time, technical expertise, and cost .

Due to advances in technology of enteral feeding tubes and delivery systems, specialization of health professionals, and better education of parents and caregivers, the administration of enteral nutrition has been associated with improved clinical outcome and safety profiles. Enteral nutrition therapy is easier and safer to administer than is par-enteral nutrition. Not only are the risks of intravenous access avoided, but there is also a wider margin for error with most metabolic complications. As a result, enteral nutrition therapy is easier to administer in low-intensity hospitals and patient care settings, including the home. However, compared with normal diet, tube feedings require extra time and effort to administer and this additional care need may contribute to increased burden and stress for families and caregivers .

This study was designed as a randomized controlled trial to compare the effect of intermittent enteral feeding by using syringe pump versus hospital blended feeding by using feeding bag on the nutritional status and complications among ICU patients.

Methods Design Structured as a randomized-controlled prospective study, the objective of this study was to compare the efficacy of intermittent enteral feeding by using syringe pump versus hospital blended formula by using feeding bag on reducing complications and improving the nutritional status of patients the intensive care units.

Setting Data was collected from assiut university hospitals .

Sample The study population consisted of patients eighteen to sixty years old, hospitalized and treated in critical and trauma intensive care units. The inclusion criteria stipulated that the patient was between eighteen and sixty years old; both genders were included; patients with a functional gastrointestinal tract and poor oral nutritional intake and agreed to participate in the study. A power calculation estimated that in order to detect an effect size of 11.8 difference in mean of protein level between the two studied groups, with a p-value < 0.05 and 80% power, confidence level 0.95, a sample size of 22 patients for each group was needed. However, 60 patients were attempted in this research work to avoid non-response rate (30 for each group). This calculated using G Power 3.1 . The study data was collected between June 2019 and December 2019.

Instruments and measurements Three tools used in this study were developed by the researcher based on reviewing of the literature. The first tool was general assessment sheet used to monitor hemodynamic parameters included (Mean arterial pressure (MAP) taken from bed side monitor, heart rate (HR), temperature, respiratory rate and CVP readings, physical examination done every day and included neurological examination and chest examination regarding disturbances, chest x-ray assessment, mode of ventilation and duration of mechanical ventilation, fluid balance assessment., assessment of laboratory findings in addition to socio-demographic and medical data.

The second tool is feeding assessment sheet was developed by the researcher and used to assess BMI after assessing height and weight; assessment of amount of water, protein, calories was given per day; assessment of mode of enteral feeding ; residual volume assessment; period of feeding rest and frequency .

The third tool is Patients' outcomes evaluation sheet which was developed by the researcher and used to assess patients' outcomes and complications . .

Intervention After getting ethical clearance patients were enrolled in the study, patients were selected based on the inclusion and exclusion criteria. Following an initial assessment, the patients were assigned to one of the two groups by block randomization.

Both groups received 3000 ml of feed per day and the same formula per day which was 30-35 ml/kg of water, 0.8 g/kg of protein and 2000 k cal of calories for females and 2500 K cal for males. The only manipulation was in the flow rate and the device which the feed was administered.

Intermittent enteral feeding group received intermittent feeding as the feed was given over a 24 hour period with intervals of rest (e.g. three hours feeding two hours rest) by using syringe pump and Feeds were administered according to guidelines as the head of the patient's bed was elevated at least 30 degrees from the horizontal before initiating feeding, the feeding schedule was started at a rate of 50 ml/hr in adults to promote tolerance,the administration rate of isotonic formulas increased in 20-25 ml/hr increments every eight hours until the desired rate was achieved, the tube was flushed regularly with 20 to 30 ml of warm water every four hours during continuous feeding and before and after intermittent feeding and medication administration, the gastric residual volume was checked every 4-6 hr routinely Feeding bag group received hospital blended formula which was 300 ml of feeds every 24 hrs with 4 hrs rest at night and given in 10 minutes with following the same guidelines in the intermittent enteral feeding group.

Data collection The data were collected from the first day of admission after stabilization of the patient's condition and extended to 7 days, every day then the data were recorded in the developed tools.The researcher assigned study sample (30 patients) to two groups (intermittent enteral feeding group, feeding bag group).

For intermittent enteral feeding group: The researcher assessed patients who were receiving intermittent enteral feeding. For feeding bag group: The researcher assessed patients who received hospital blended formula.

Ethical considerations Approval for the study was obtained from the Ethics Committee of the faculty of nursing with no risk for study subject during application of the study as the study followed common ethical principles in clinical research and written consent was obtained from patients or guidance that participated in the study after explaining the nature and purpose of the study.

Patient was assured that the data of this research was not be reused without second permission, confidentiality and anonymity was assured and the patients had the right to refuse to participate or withdraw from the study without any rational at any time.

.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* patients of both genders.
* patients with a functional gastrointestinal tract and poor oral nutritional intake.

Exclusion Criteria:

* patients for whom par-enteral nutrition would be more suitable.
* patients wit GIT obstruction or fistula.
* patients with ischemic bowel.
* patients in whom enteral feeding access is not available

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
change in serum protein level | for 10 days
  by using serum protein test which will be assessed daily, there will be change in the serum protein level to the normal value
change in the rate of complications | for 10 days
  by using evaluation outcomes tool , complications will be assessed 3 times through the study

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Mohamed, Principal Investigator — Assiut University
Locations (1):
- Faculty of Nursing, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No